CLINICAL TRIAL: NCT04027283
Title: Acute Effects of the Two Alternative Sweeteners D-allulose and Erythritol on Gastrointestinal Hormone Secretion and Glycemic Control
Brief Title: Acute Effects of the Two Alternative Sweeteners D-allulose and Erythritol on Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: PolyAlluLac
Record Dates: First submitted 2019-07-02; First posted 2019-07-19 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Physiological Satiation Mechanisms
MeSH Terms: interventions — Erythritol; lactisole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Erythritol (Active Comparator): 18 volunteers receive 50g erythritol dissolved in 300mL tap water via a nasogastric tube
  Interventions: Dietary Supplement: Erythritol
- Erythritol + lactisole (Active Comparator): 18 volunteers receive 50g erythritol with lactisol (450ppm) dissolved in 300mL tap water via a nasogastric tube
  Interventions: Dietary Supplement: Erythritol + lactisole
- D-allulose (Active Comparator): 18 volunteers receive 25g D-allulose dissolved in 300mL tap water via a nasogastric tube
  Interventions: Dietary Supplement: D-allulose
- D-allulose + lactisole (Active Comparator): 18 volunteers receive 25g D-allulose with lactisole (450ppm) dissolved in 300mL tap water via a nasogastric tube
  Interventions: Dietary Supplement: D-allulose + lactisole
- Tap water (Placebo Comparator): 18 volunteers receive 300mL tap water via a nasogastric tube
  Interventions: Dietary Supplement: Tap water
- Tap water + lactisole (Placebo Comparator): 18 volunteers receive 300mL tap water + lactisole (450ppm) via a nasogastric tube
  Interventions: Dietary Supplement: Tap water + lactisole

INTERVENTIONS:
Dietary Supplement: Erythritol — 50g erythritol dissolved in 300mL tap water
  Other Names: E968-Erythritol
  Arms: Erythritol
Dietary Supplement: Erythritol + lactisole — 50g erythritol + lactisole (450ppm) dissolved in 300mL tap water
  Other Names: E968-Erythritol
  Arms: Erythritol + lactisole
Dietary Supplement: D-allulose — 25g D-allulose dissolved in 300mL tap water
  Arms: D-allulose
Dietary Supplement: D-allulose + lactisole — 25g D-allulose + lactisole (450ppm) dissolved in 300mL tap water
  Arms: D-allulose + lactisole
Dietary Supplement: Tap water — 300mL tap water
  Arms: Tap water
Dietary Supplement: Tap water + lactisole — 300mL tap water + lactisole (450ppm)
  Arms: Tap water + lactisole

SUMMARY:
The aim of this project is to investigate the effect of intragastric (ig) D-allulose on metabolic parameters in general and to investigate the effect of sweet taste receptor blockade on GI hormone responses, glycemic control, gastric emptying (GE) rates and appetite-related sensations to ig administration of erythritol and D-allulose.

DETAILED DESCRIPTION:
Erythritol (natural non-caloric sweetener) could be an ideal candidate substitute for sugar as it may reduce caloric intake without compensatory overeating or earlier return of hunger. Moreover, it may serve as a physiological tool to disentangle the effects of gastrointestinal (GI) sweet taste receptor stimulation, (an)orexigenic hormone secretion, and glucose metabolism/caloric content on food intake regulation in vivo in humans. However, its effects on appetite, satiation, and satiety have not been studied systematically. Moreover, the mechanisms underlying erythritol-induced anorexigenic GI hormone release have not been investigated so far.

D-allulose is a sugar substitute with almost zero calories and is naturally occurring in small quantities. Apart from its use as sugar replacement, D-allulose seems to favorably affect glycemic control and metabolism as could be shown in animal trials and in a few human trials. However, to date the effects of D-allulose on GI hormone secretion, appetite-related sensations and glycemic control, are not or insufficiently studied in humans.

The aim of this project is therefore to investigate the effect of intragastric (ig) D-allulose on metabolic parameters in general and to investigate the effect of sweet taste receptor blockade on GI hormone responses, glycemic control, gastric emptying (GE) rates and appetite-related sensations to ig administration of erythritol and D-allulose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy normal weight subjects with a body-mass index of 19.0-24.9
* Normal eating habits (no diets; no dietary changes)
* Age 18-55 years
* Stable body weight for at least three months
* Informed Consent as documented by signature (Appendix Informed Consent Form)

Exclusion Criteria:

* Pre-existing consumption of erythritol or D-allulose on a regular basis (usage of erythritol or D-allulose as sugar replacement; in contrast, erythritol-containing toothpaste is allowed)
* Substance abuse
* Regular intake of medications, except anticonceptives
* Chronic or clinically relevant acute infections
* Pregnancy: although no contraindication, pregnancy might influence metabolic state. Women who are pregnant or have the intention to become pregnant during the course of the study are excluded. In female participants a urine pregnancy test is carried out upon screening.
* Participation in another study with investigational drug within the 30 days preceding and during the present study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Effects on GI hormone response - GLP-1 | Changes from baseline to three hours after treatment. Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 120, and 180minutes (after administration).
  Plasma GLP-1 will be measured with a commercially available immunoassay kit (MILLIPLEX® MAP; Millipore Corporation, Billerica, MA, USA).
Effects on GI hormone response - PYY | Changes from baseline to three hours after treatment. Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 120, and 180minutes (after administration).
  Plasma PYY, and ghrelin will be measured with a commercially available immunoassay kit (MILLIPLEX® MAP; Millipore Corporation, Billerica, MA, USA).
Effects on GI hormone response - ghrelin | Changes from baseline to three hours after treatment. Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 120, and 180minutes (after administration).
  Plasma ghrelin will be measured with a commercially available immunoassay kit (MILLIPLEX® MAP; Millipore Corporation, Billerica, MA, USA).
Effects on GI hormone response - CCK | Changes from baseline to three hours after treatment. Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 120, and 180minutes (after administration).
  Plasma cholecystokinin (CCK) levels will be measured with a sensitive radioimmunoassay using a highly specific antiserum.
Effects on GI hormone response - motilin | Changes from baseline to three hours after treatment. Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 120, and 180minutes (after administration).
  Plasma motilin levels will be measured with a sensitive radioimmunoassay as previously described using 125I [Nle13] human motilin as tracer and rabbit anti-human Nle13 motilin antibody (final dilution 1/12000).

SECONDARY OUTCOMES:
Effects on glycemic control - plasma glucose | Changes from baseline to three hours after treatment. Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 120, and 180minutes (after administration).
  Blood glucose concentrations will be measured by a commercial hexokinase-glucose-6-phosphate-dehydrogenase method (Roche, Basel, Switzerland).
  Insulin, c-peptide and glucagon will be measured with a commercially available immunoassay kit (MILLIPLEX® MAP; Millipore Corporation, Billerica, MA, USA). The lowest level of insulin that can be detected by this assay is 87 pg/mL when using a 25 µL sample. The lowest level of c-peptide that can be detected by this assay is 9.5 pg/mL when using a 25 µL sample. The lowest level of glucagon that can be detected by this assay is 13 pg/mL when using a 25 µL sample. The intra-assay coefficient of variation for all peptides (insulin, c-peptide and glucagon) is below 10%, whereas the inter-assay coefficient of variation is below 15%.
Effects on glycemic control - plasma insulin | Changes from baseline to three hours after treatment. Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 120, and 180minutes (after administration).
  Insulin will be measured with a commercially available immunoassay kit (MILLIPLEX® MAP; Millipore Corporation, Billerica, MA, USA). The lowest level of insulin that can be detected by this assay is 87 pg/mL when using a 25 µL sample. The intra-assay coefficient of variation for insulin is below 10%, whereas the inter-assay coefficient of variation is below 15%.
Effects on glycemic control - plasma c-peptide | Changes from baseline to three hours after treatment. Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 120, and 180minutes (after administration).
  C-peptide will be measured with a commercially available immunoassay kit (MILLIPLEX® MAP; Millipore Corporation, Billerica, MA, USA). The lowest level of c-peptide that can be detected by this assay is 9.5 pg/mL when using a 25 µL sample. The intra-assay coefficient of variation for c-peptide is below 10%, whereas the inter-assay coefficient of variation is below 15%.
Effects on glycemic control - plasma glucagon | Changes from baseline to three hours after treatment. Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 120, and 180minutes (after administration).
  Glucagon will be measured with a commercially available immunoassay kit (MILLIPLEX® MAP; Millipore Corporation, Billerica, MA, USA). The lowest level of glucagon that can be detected by this assay is 13 pg/mL when using a 25 µL sample. The intra-assay coefficient of variation for glucagon is below 10%, whereas the inter-assay coefficient of variation is below 15%.
Effects on gastric emptying rate | Changes from baseline to four hours after treatment. Breath samples will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 75, 90, 105, 120, 150, 180 and 240minutes (after administration).
  Gastric emptying rate will be determined using a 13C-sodium acetate breath test.
Effects on blood lipids | Changes from baseline to two hours after treatment. Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 30, 60, and 120minutes (after administration).
  Analyses of blood lipids are carried out in the hospital laboratory.
Effects on uric acid | Changes from baseline to two hours after treatment. Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 30, 60, and 120minutes (after administration).
  Analyses of uric acid are carried out in the hospital laboratory.
Effects on hsCRP (high sensitive c-reactive protein) | Changes from baseline to two hours after treatment. Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 30, 60, and 120minutes (after administration).
  Analyses of hsCRP are carried out in the hospital laboratory.
Effects on appetite-related sensations | Changes from baseline to four hours after treatment. Visual analogue scales will be recorded at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 75, 90, 105, 120, 150, 180 and 240minutes (after administration).
  Appetite perceptions (feelings of: a) hunger, b) satiety) are assessed by visual analogue scale (VAS). Visual analogue scales consist of a horizontal, unstructured, 10-cm line representing the minimum (0.0 points) to the maximum rating (10.0 points). Subjects assign a vertical mark across the line to indicate the magnitude of their subjective sensation at the present time point. The measurement is quantified by the distance from the left end of the line (minimum rating) to the subject's vertical mark.

OTHER OUTCOMES:
Effects on GI tolerance | Changes from baseline to four hours after treatment. GI tolerance will be recorded at time=-10, time=30, time=60, time=90, time=120, time=150, time=180, and time=240minutes.
  GI symptoms will be assessed by use of a checklist including the following questions: abdominal pain, nausea, vomiting, diarrhoea, borborygmi, abdominal distension, eructation and increased flatus.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Christin Meyer-Gerspach, PD, PhD, Principal Investigator — St. Clara Research Ltd.
Locations (1):
- St. Claraspital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No